CLINICAL TRIAL: NCT02670668
Title: Single Centre，Exploratory，Parallel and Retrospective Study to Analysis the Mutation and Expression of BRCA1/2 and Other Potential Genes in Triple-negative Breast Cancer
Brief Title: Mutation of BRCA1/2 and Other Potential Genes in Triple-negative Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, A-Yong Cao, MD, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ESR-14-10562
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: BRCA1/2;Mutations;Neoadjuvant chemotherapy;TNBC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mutation analysis- NACwith PCR (Experimental): consisting of 50 patients undergoing NACwith pathological compete response
  Interventions: Other: Mutation analysis
- Mutation analysis-NAC with SD/PD. (Experimental): consisting of 50 patients undergoing NAC with SD/PD
  Interventions: Other: Mutation analysis

INTERVENTIONS:
Other: Mutation analysis

SUMMARY:
The study is to determine the prevalence of potential chemo-response related genes mutation in TNBC patients between pCR and SD/PD group, which achieved after NAC; and to evaluate potential relationship between these gene mutations and NAC-response in TNBC patients.Based on the results,we can further characterize TNBC from a phenotypical and molecular perspective, in order to identify potential new target agents and to individualize the treatment.

DETAILED DESCRIPTION:
This is single centre，exploratory，parallel and retrospective study to analysis the mutation and expression of tBRCA1/2 and other potential genes in triple-negative breast cancer. Patients received neoadjuvant chemotherapy with paclitaxel and carboplation are enrolled in this study. The participants are required to have clinical stage II or III breast cancer with a clinical or radiographically measurable residual tumor after core biopsy. We will enroll the patients of pCR or SD/PD, which achieved after complete NAC. Every group will enroll 50 patients. This study is to identify relationship between different gene mutations and expression, which may be targeted with currently available investigational drugs, and chemo-response.

Patients who will fulfil all inclusion/exclusion criteria. We conducted a retrospective chart review of the 100 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving neoadjuvant chemotherapy with paclitaxel and carboplation are enrolled in this study.

* (1) histologically confirmed mainly invasive breast carcinoma
* (2) a unilateral and non-inflammatory tumors
* (3) status of ER, PR and HER-2 are available and negative
* (4) The participants are required to have clinical stage II or III breast cancer with a clinical or radiographically measurable residual tumor after core biopsy.
* (5)patients had pathological evaluation after NAC
* (6) the pathologic tissues are available for immunohistochemistry and next generation sequencing

Exclusion Criteria:

* (1) carcinoma in situ
* (2) received less than 4 cycles neoadjuvant chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Gene mutation prevalence of tBRCA1/2, HRR, or other chemo-response related genes in TNBC patients between pCR and SD/PD, which achieved after NAC | Baseline

SECONDARY OUTCOMES:
To evaluate potential relationship between these gene mutations and NAC-response in TNBC patients | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ayong Cao, MD, Principal Investigator — Fudan University
Locations (1):
- Department of Breast Surgery, Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided